CLINICAL TRIAL: NCT03325452
Title: A Pilot Study Evaluating the PROgnostic Contribution of Venous Lactate for the Recovery of Spontaneous Cardiac Activity, Following an Extra-hospital Cardiac Arrest "PROLAC Study"
Brief Title: Evaluating Prognostic Contribution of Lactate on Recovery of Spontaneous Cardiac Activity After Cardiac Arrest
Acronym: PROLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-AOI-03
Record Dates: First submitted 2017-10-23; First posted 2017-10-30 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Cardio-respiratory Arrest, Prolactin
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: The hypothesis of our study is that the evaluation of the initial lactate in the early cardiopulmonary resuscitation could be a prognostic factor of RACS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardio-respiratory arrest (Experimental)
  Interventions: Biological: venous lactate

INTERVENTIONS:
Biological: venous lactate — value of venous lactate

SUMMARY:
Incidence of non-hospital cardio-respiratory arrest (ACR) in France is around 40 000 cases per year, with mortality remaining very high, with 75% of patients dying before arrival in hospital. The investigators know some validated predictive factors for recovery of spontaneous cardiac activity (RACS) such as age, no flow (time between ACR and onset of CPR), type of initial electrical activity (FV, TVSP), or the value of CO2 expired.

However, the use of these prognostic criteria in the conduct of CPR maneuvering is in practice limited. Lactate is now a well-known prognostic biological marker used in many pathological conditions such as shock states or the severe traumatized patient. Some data have also demonstrated the prognostic value of lactate on morbidity and mortality after ACR after resumption of spontaneous cardiac activity.

The hypothesis of our study is that the evaluation of the initial lactate in the early cardiopulmonary resuscitation could be a prognostic factor of RACS.

DETAILED DESCRIPTION:
Incidence of non-hospital cardio-respiratory arrest (ACR) in France is around 40 000 cases per year, with mortality remaining very high, with 75% of patients dying before arrival in hospital. This disease is associated with a high morbidity since today the investigator find less than 5% survival at 1 year with a favorable neurological outcome.

The recommendations of ILCOR 2015 underline in this case the importance of implementing therapeutic measures in the extra-hospital step. Indeed, the survival of ACR patients will depend mainly on the alert delay at the UAS center, the immediate implementation of cardiopulmonary resuscitation (CPR) maneuvers and the early delivery of external electric shock.

The investigators know some validated predictive factors for recovery of spontaneous cardiac activity (RACS) such as age, no flow (time between ACR and onset of CPR), type of initial electrical activity (FV, TVSP), or the value of CO2 expired.

However, the use of these prognostic criteria in the conduct of CPR maneuvering is in practice limited.

Today, none of these prognostic factors allow us to adapt the cardiopulmonary resuscitation maneuvers to the different clinical situations, and it is recognized that a CPR must be carried out for 30 minutes in all cases.

On the basis of these data, it seemed important to investigate other predictive factors for RACS, which would remain simple to implement, and allow case-by-case customization the cardiopulmonary resuscitation.

Lactate is now a well-known prognostic biological marker used in many pathological conditions such as shock states or the severe traumatized patient. Some data have also demonstrated the prognostic value of lactate on morbidity and mortality after ACR after resumption of spontaneous cardiac activity. Unfortunately, all of these studies were carried out intra-hospital. To date, no prospective study has demonstrated the prognostic value of a lactate assay as soon as the pre-hospital medical team arrives and during pre-hospital cardiopulmonary resuscitation.

An experimental study published in the American Journal of Emergency Medicine in 1985, however, suggests that early evaluation of lactate in the course of cardiac arrest may be a valuable prognostic factor. Indeed, in this study on canine cardiac arrest experimental model, Donna et al found that the lactate concentration would reliably predict the no-flow describing an linear increase of lactate as a function of the no-flow duration. If these results can be extrapolated to humans, lactate measurement from the arrival of the pre-hospital medical team could provide an estimate of the no-flow period and therefore a reliable and easily reproducible predictive factor for RACS .

In addition, improvements in biomedical equipment allow us to perform lactate assays directly at the patient's bedside, with reliable results in just 13 seconds.

The hypothesis of our study is that the evaluation of the initial lactate in the early cardiopulmonary resuscitation could be a prognostic factor of RACS.

For this purpose, the investigators propose to carry out a prospective, open, multicenter intervention study in different SMURs in the PACA region, in France.

ELIGIBILITY:
Inclusion Criteria:

* Male >18 years of age
* Women over 50 years of age (ie, with amenorrhea> 1 year).
* Victim of non-traumatic cardiopulmonary arrest.
* Medical decision to start or continue cardiopulmonary resuscitation.
* Consent of family or person of trust if present (and patient as soon as possible).
* patient affiliated to the social security

Exclusion Criteria:

* Refusal of family or trusted person to participate in the study
* Pre-paramedical management with use of adrenaline and protection of the airways
* Use of the intraosseous line from the outset or after failure of the peripheral venous pathway by the medical team outside hospital
* Minor Patient
* vulnerable patient under legal protection (guardianship or curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
venous lactate | at baseline
  The main evaluation criteria will be the value of the venous lactate that was measured during insertion of the peripheral venous line at the arrival of the medical team (= T0) in patients in cardiac arrest

SECONDARY OUTCOMES:
Initial value of capillary lactate | at baseline
  to compare with the initial venous lactate value measured at the peripheral venous laying
The no-flow | at baseline
  This data will be obtained by interrogating the witnesses present during the cardiac arrest.
The kinetics of capillary lactate | at time = 10 minutes
  to evaluate by the variability of capillary lactate levels
The kinetics of capillary lactate | at time = 20 minutes
  to evaluate by the variability of capillary lactate levels
The kinetics of capillary lactate | at time = 30 minutes
  to evaluate by the variability of capillary lactate levels

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Provences Alpes Cote d'Azur, France